CLINICAL TRIAL: NCT03333486
Title: A Phase II Trial of Haploidentical Allogeneic Stem Cell Transplantation Utilizing Mobilized Peripheral Blood Stem Cells
Brief Title: Fludarabine Phosphate, Cyclophosphamide, Total Body Irradiation, and Donor Stem Cell Transplant in Treating Patients With Blood Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility analysis determined closure
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 40916; NCI-2017-01949 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 40916 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Leukemia in Remission; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Acute Myeloid Leukemia With FLT3/ITD Mutation; Acute Myeloid Leukemia With Gene Mutations; Aplastic Anemia; B-Cell Non-Hodgkin Lymphoma; CD40 Ligand Deficiency; Chronic Granulomatous Disease; Chronic Leukemia in Remission; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Congenital Amegakaryocytic Thrombocytopenia; Congenital Neutropenia; Congenital Pure Red Cell Aplasia; Glanzmann Thrombasthenia; Immunodeficiency Syndrome; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Paroxysmal Nocturnal Hemoglobinuria; Plasma Cell Myeloma; Polycythemia Vera; Recurrent Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome; Severe Aplastic Anemia; Shwachman-Diamond Syndrome; Sickle Cell Disease; T-Cell Non-Hodgkin Lymphoma; Thalassemia; Waldenstrom Macroglobulinemia; Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Aplastic; Lymphoma, B-Cell; Granulomatous Disease, Chronic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Congenital amegakaryocytic thrombocytopenia; Neutropenia, Severe Congenital, Autosomal Recessive 3; Anemia, Diamond-Blackfan; Thrombasthenia; Immunologic Deficiency Syndromes; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Hemoglobinuria, Paroxysmal; Multiple Myeloma; Polycythemia Vera; Lymphoma, Non-Hodgkin; Shwachman-Diamond Syndrome; Anemia, Sickle Cell; Lymphoma, T-Cell; Thalassemia; Waldenstrom Macroglobulinemia; Wiskott-Aldrich Syndrome | interventions — Cyclophosphamide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (fludarabine, cyclophosphamide, TBI, PBSCT) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 2 hours on days -6 and -5. Patients undergo TBI on days -1 and PBSCT on day 0.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; peripheral stem cell support; Peripheral Stem Cell Transplant; peripheral stem cell transplantation
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well fludarabine phosphate, cyclophosphamide, total body irradiation, and donor stem cell transplant work in treating patients with blood cancer. Drugs used in chemotherapy, such as fludarabine phosphate and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient?s immune cells and help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the rate of relapse, defined as recurrence of underlying disease or progression of underlying disease, at 1 year in patients who receive haploidentical peripheral blood stem cells (PBSCs) after reduced intensity conditioning and post-transplant cyclophosphamide and tocilizumab (or tocilizumab alternative).

SECONDARY OBJECTIVES:

I. To evaluate safety including development of acute graft versus host disease (GVHD) and death at 100 days post-transplant, as well as other treatment related toxicities including chronic GVHD, engraftment rate, non-relapse mortality, progression free survival (PFS) at one year, and overall survival (OS) at one year, as compared with historical controls.

TERTIARY OBJECTIVES:

I. Correlative studies will include chimerism analysis by molecular analysis and evaluation of immune reconstitution by cytomegalovirus (CMV) dextramer analysis using flow cytometry.

OUTLINE:

Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -6 to -2 and cyclophosphamide IV over 2 hours on days -6 and -5. Patients undergo total body irradiation (TBI) on days -1 and peripheral blood stem cell transplantation (PBSCT) on day 0.

After completion of study treatment, patients are followed up at 30 and 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Any disease that is considered transplant eligible per TCT standards
* Disease response noted (i.e. CR, non-CR, or not applicable): Assessed as per disease specific criteria
* Suitable related haploidentical donor identified per transplant service:

  * Recipient should not have HLA antibodies to potential donor. If the recipient does have HLA antibodies to the potential donor, an alternative donor is preferred; however, if there are no suitable alternative donors, the anti-HLAt antibodies should be depleted per transplant service guidelines.
  * Haploidentical donors that are ABO compatible with the recipient are preferred. Minor ABO incompatibility is preferred to major ABO incompatibility. Major ABO incompatibility between recipient and donor is the least preferred but still acceptable for this study.
  * It is preferred that the haploidentical donor must be available to donate on day -1 and day 0, so that fresh product can be processed by the Stem Cell lab and administered to the patient on day 0.While less preferable, cryopreserved product may be utilized with this product.
* Diffusing capacity of the lung for carbon monoxide (DLCO) > 40% predicted, corrected for hemoglobin and/or alveolar ventilation
* Left ventricular ejection fraction > 40%
* Bilirubin, liver alkaline phosphatase, serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) =< 3 x upper limit of normal
* Calculated creatinine clearance > 40 cc/min by the modified Cockcroft-Gault formula for adults or the Schwartz formula for pediatrics
* Have a Karnofsky (adult) or Lansky (for =< 16 years) performance status >= 60%
* Patient must be able to pass radiation evaluation (i.e.: able to receive 200 cGy)
* Patients who have failed a prior autologous transplant are eligible; however, at least 90 days must have elapsed between the start of this reduced intensity conditioning regimen and the last transplant if patient had a prior autologous BMT
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an independent ethics committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* If patient is planned to use a fully matched donor, patient is excluded from trial; patient must be planned to undergo a haploidentical matched transplant to participate on study. Patient is still eligible for trial regardless of donor options if PI feels that haplo transplant is in the patient's best interest per clinical decision
* Exclusion Criteria:
* Participants who have had chemotherapy (not including molecularly targeted agents; examples include, but are not limited to, tyrosine kinase inhibitors such as FLT3 inhibitors and IDH2 inhibitors), radiation treatment and/or surgery 7 days prior to starting conditioning regimen. Those who have not recovered sufficiently from adverse events due to agents administered more than 2 weeks earlier are also ineligible. Exceptions may be made on a case-by-case basis after discussion with the PI
* Uncontrolled central nervous system (CNS) disease (for hematologic malignancies) Per PI discretion
* Child-Pugh class B and C liver failure
* Concomitant active malignancy that would be expected to require chemotherapy within 3 years of transplant (other than non-melanoma skin cancer) Exception would include any concurrently existing malignancy that could be treated with a transplant per PI discretion (Example: Patient has AML but a history of mastocytosis)
* Patients who have received maximally allowed doses (given in 2 Gy fractionations, or equivalent) of previous radiation therapy to various organs; patients who previously have received a higher than allowed dose of radiation to a small lung, liver and brain volume, will be evaluated by the radiation oncologist to determine if the patient is eligible for study
* Uncontrolled diabetes mellitus, cardiovascular disease, active serious infection or other condition which, in the opinion of treating physician, would make this protocol unreasonably hazardous for the patient
* Known human immunodeficiency virus (HIV) positive
* Pregnant or nursing female participants
* Patients who in the opinion of the treating physician are unlikely to comply with the restrictions of allogeneic stem cell transplantation based on formal psychosocial screening
* Patients with donor specific HLA antibodies with a titer greater than 3000 MFI (whether or not they have undergone a desensitization protocol)
* Patients who have undergone a prior allogeneic hematopoietic or (other organ) transplant
* Treating physician considers the potential HLA haploidentical donor to be ineligible to receive G-CSF, and/or concern on the part of the treating physician for risk of harm to the potential donor with administration of G-CSF, and/or refusal by the potential donor (or donor's guardian) to receive G-CSF
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Received an investigational agent within 14 days prior to enrollment. Exceptions may be made on a case-by-case basis after discussion with PI

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip McCarthy, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Started | 31
Completed | 29
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Relapse Rate
Description: The number of participants that relapse within 1 year.
Time Frame: At 1 year
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
Participants | 14

2. Secondary Outcome: ANC Engraftment Rate, the Percentage of Participants That Had a Successful Engraftment
Description: Absolute Neutrophil Count Engraftment rate was defined as the number of participants that received an engraftment within 1 year post-transplant and ANC > 0.5x10^9/L for three consecutive days, out of the total number of participants. The rate was computed with corresponding exact 95% confidence intervals based on the methodology of Clopper and Pearson.
Time Frame: At 1 year post-transplant
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
percentage of participants | 84 [66.0 to 95.0]

3. Secondary Outcome: Platelet Engraftment Rate, the Percentage of Participants That Had a Successful Engraftment
Description: Platelet Engraftment rate was defined as the number of participants that received an engraftment within 1 year post-transplant and the platelets >= 20 x 10^9/L after 7 consecutive days with no platelet transfusions, out of the total number of participants. The rate was computed with corresponding exact 95% confidence intervals based on the methodology of Clopper and Pearson.
Time Frame: At 1 year post-transplant
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
percentage of participants | 77 [59 to 90]

4. Secondary Outcome: Proportion of Participants With Acute Graft Versus Host Disease (GVHD)
Description: Will be computed with corresponding exact 95% confidence intervals based on the methodology of Clopper and Pearson.
Time Frame: At 100 days post-transplant
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
proportion of participants | 0.3226 [0.1668 to 0.5137]

5. Secondary Outcome: Proportion of Participants With Chronic Graft Versus Host Disease (GVHD)
Description: Will be computed with corresponding exact 95% confidence intervals based on the methodology of Clopper and Pearson.
Time Frame: At 1 year post-transplant
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
proportion of participants | 0.1935 [0.0745 to 0.3747]

6. Secondary Outcome: Overall Survival
Description: Will be computed with corresponding exact 95% confidence intervals based on the methodology of Clopper and Pearson. Will be obtained using the product-limit based Kaplan-Meier method.
Time Frame: up to 5 years and 8 months
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
months | 15.7 [7.1 to NA] — Upper limit not reached

7. Secondary Outcome: Progression Free Survival
Description: as for outcome 6
Time Frame: up to 5 years and 8 months
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
months | 15.7 [5.5 to 49.5]

8. Secondary Outcome: Transplant Related Mortality
Description: Will be computed with corresponding exact 95% confidence intervals based on the methodology of Clopper and Pearson.
Time Frame: At 1 year post-transplant
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 31
proportion of participants | 0.0323 [0.0008 to 0.1670]

9. Other Pre Specified Outcome: Immune Reconstitution
Description: Will be assessed by bone marrow transplantation SOC immunophenotyping panel and by analysis of cytomegalovirus-specific immunity.
Time Frame: Up to 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Lymphoid Chimerism Expressed as a Percentage of Donor Cells
Description: Mean lymphoid chimerism expressed as a percentage of donor cells
Time Frame: At 30 days
Population: All treated and eligible patients. Samples were not obtained at day 100 for 8 subjects.
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 23
percentage of donor cells | 99.85 (0.46)

11. Other Pre Specified Outcome: Myeloid Chimerism Expressed as a Percentage of Donor Cells
Description: Mean myeloid chimerism expressed as a percentage of donor cells
Time Frame: At 100 days
Population: All treated and eligible patients. Samples were not obtained at day 100 for 8 subjects.
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
Number analyzed (Participants) | 23
percentage of donor cells | 99.93 (0.22)

ADVERSE EVENTS:
Time Frame: 5 years and 8.5 months
Arm/Group | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT)
All-Cause Mortality (participants affected / at risk) | 17/31
Serious Adverse Events (participants affected / at risk) | 8/31
Other Adverse Events (participants affected / at risk) | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT) (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (3)
Lung infection (Infections and infestations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Fludarabine, Cyclophosphamide, TBI, PBSCT) (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (15)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 17 (22)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 18 (20)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (11)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Edema face (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (12)
Fever (General disorders) | 5 (5)
Flu like symptoms (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 10 (12)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 7 (8)
Infections and infestations - Other, specify (Infections and infestations) | 7 (10)
Otitis media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 6 (6)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (4)
Presyncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT03333486/Prot_SAP_000.pdf